CLINICAL TRIAL: NCT07375446
Title: Efficacy and Safety of a Traditional Chinese Medicine Hand-Foot Soak for Chemotherapy-Induced Peripheral Neuropathy and Hand-Foot Syndrome
Brief Title: Traditional Chinese Medicine Hand-Foot Soak for Chemotherapy-Induced Peripheral Neuropathy and Hand-Foot Syndrome
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M20250937
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Patients With Solid Tumors
Keywords: traditional Chinese medicine (TCM), chemotherapy-induced peripheral neuropathy (CIPN), hand-foot syndrome (HFS)
MeSH Terms: conditions — Hand-Foot Syndrome | interventions — Medicine, Chinese Traditional

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Traditional Chinese medicine group: Patients received a topical TCM treatment. The formula consisted of: Ramulus Cinnamomi (Guizhi), Radix Angelicae Sinensis (Danggui) , Radix Aconiti Lateralis Preparata (Zhi Chuanwu) , Caulis Spatholobi (Jixueteng), Rhizoma Chuanxiong (Chuanxiong) , Radix Astragali (Huangqi), Rhizoma Dioscoreae Nipponicae (Chuanshanlong) , Herba Speranskiae Tuberculatae (Tougucao), Radix Paeoniae Rubra (Chishao), and Radix Sophorae Flavescentis (Kushen Pian).
  The herbs were decocted in 1000-2000ml of 37-41℃ water. Patients were instructed to soak their hands and feet in the warm solution for 20-30 minutes twice daily.
  Interventions: Drug: Traditional Chinese Medicine

INTERVENTIONS:
Drug: Traditional Chinese Medicine — Ramulus Cinnamomi (Guizhi) , Radix Angelicae Sinensis (Danggui) , Radix Aconiti Lateralis Preparata (Zhi Chuanwu), Caulis Spatholobi (Jixueteng) , Rhizoma Chuanxiong (Chuanxiong) , Radix Astragali (Huangqi) , Rhizoma Dioscoreae Nipponicae (Chuanshanlong) , Herba Speranskiae Tuberculatae (Tougucao) , Radix Paeoniae Rubra (Chishao) , and Radix Sophorae Flavescentis (Kushen Pian)

SUMMARY:
Systemic therapies, including chemotherapy, targeted therapy, and immunotherapy, are cornerstones of modern oncology and have significantly extended patient survival. However, these treatments are frequently associated with adverse reactions that can impair patients' quality of life. Among the most common and debilitating are chemotherapy-induced peripheral neuropathy (CIPN) and hand-foot syndrome (HFS).

Currently, no universally effective standard of care exists for either CIPN or HFS. Interventions such as duloxetine for CIPN or empirical vitamin use for HFS offer limited efficacy and are not robustly supported by evidence. This unmet clinical need has driven interest in complementary approaches. In recent years, traditional Chinese medicine (TCM) has been rigorously evaluated in high-quality clinical trials for various conditions, showing benefits in cardiovascular disease and oncology. However, while some studies have explored systemic TCM for preventing CIPN, research on topical TCM therapies for established CIPN and HFS is scarce. We therefore conducted this retrospective study to investigate the efficacy and safety of a topical TCM hand-foot soak for these conditions, using patient-reported outcome measures to assess its impact on symptoms and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* (1) The patient is over 18 years old, with no gender restrictions; (2) Pathology confirmed malignant tumor, including digestive tract tumor, lung cancer, breast cancer, etc; (3) Received systemic anti-tumor treatment, including chemotherapy, targeted therapy, etc; (4) Combination of HFS or CIPN after anti-tumor treatment; (5) After the occurrence of HFS or CIPN, according to the diagnosis and treatment routine or the patient's wishes, traditional Chinese medicine topical treatment is used, or western medicine such as methylcobalamin/vitamin B is taken orally, or no intervention measures are used; (6) The main organ functions are normal, and there are no severe abnormalities in blood, heart, lung, liver, kidney, bone marrow, or immunodeficiency diseases; (7) The time from the end of the previous use of traditional Chinese medicine and traditional Chinese patent medicines and simple preparations to the start of the study must be ≥ 2 weeks; (8) Those with good compliance can follow up on the efficacy and adverse reactions according to the requirements of the plan; (9) HFS, CIPN, and quality of life assessments were conducted before and after treatment.

Exclusion Criteria:

(1) Incomplete clinical data; (2) Before treatment, there were poor control of symptoms of diabetes peripheral neuropathy, history of nerve trauma, spinal cord compression syndrome without surgical treatment, spinal canal stenosis or spinal cord nerve root compression, central nervous system tumors; (3) Individuals with a known history of allergies to the components of this medication regimen; (4) Other situations that researchers believe are not suitable for inclusion.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: This study will enroll patients with solid tumors who received systemic anticancer therapy at the Department of Medical Oncology and Radiation Sickness, Peking University Third Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
CIPN scores | From enrollment to the end of treatment at 8 weeks"

SECONDARY OUTCOMES:
HFS Grade | From enrollment to the end of treatment at 8 weeks"

IPD SHARING:
Plan to Share IPD: Yes